CLINICAL TRIAL: NCT05139693
Title: Accuracy of Pulse Oximeters With Profound Hypoxia
Status: Completed | Type: Observational
Sponsor: Respiree Pte Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: 10-00437
Record Dates: First submitted 2021-11-17; First posted 2021-12-01 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

INTERVENTIONS:
Device: Respiree — The aim of this project is to test the accuracy of pulse oximeters during mild, moderate and severe hypoxia. This is done by comparing the reading of the pulse oximeter during brief, steady state hypoxia with a gold-standard measurement of blood oxyhemoglobin saturation (arterial blood sample processed in a laboratory hemoximeter). The data obtained is submitted by pulse oximeter manufacturers to the FDA for device approval

SUMMARY:
The aim of this project is to test the accuracy of pulse oximeters during mild, moderate and severe hypoxia. This is done by comparing the reading of the pulse oximeter during brief, steady state hypoxia with a gold-standard measurement of blood oxyhemoglobin saturation (arterial blood sample processed in a laboratory hemoximeter). The data obtained is submitted by pulse oximeter manufacturers to the FDA for device approval.

DETAILED DESCRIPTION:
The study will include at least 10 subjects (up to 14 if needed to reach the 200 necessary data points to meet the ISO 80601-2-61:2017).

Per FDA guidance, at least 2, or 15% of the subjects will have dark skin.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is male or female, aged ≥18 and <50.
2. The subject is in good general health with no evidence of any medical problems.
3. The subject is fluent in both written and spoken English.
4. The subject has provided informed consent and is willing to comply with the study procedures.

Exclusion Criteria:

1. The subject is obese (BMI>30).
2. The subject has a known history of heart disease, lung disease, kidney or liver disease.
3. Diagnosis of asthma, sleep apnea, or use of CPAP.
4. Subject has diabetes.
5. Subject has a clotting disorder.
6. The subject a hemoglobinopathy or history of anemia, per subject report or the first blood sample, that in the opinion of the investigator, would make them unsuitable for study participation.
7. The subject has any other serious systemic illness.
8. The subject is a current smoker.
9. Any injury, deformity, or abnormality at the sensor sites that in the opinion of the investigators' would interfere with the sensors working correctly.
10. The subject has a history of fainting or vasovagal response.
11. The subject has a history of sensitivity to local anesthesia.
12. The subject has a diagnosis of Raynaud's disease.
13. The subject has unacceptable collateral circulation based on exam by the investigator (Allen's test).
14. The subject is pregnant, lactating or trying to get pregnant.
15. The subject is unable or unwilling to provide informed consent, or is unable or unwilling to comply with study procedures.
16. The subject has any other condition, which in the opinion of the investigators' would make them unsuitable for the study.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study will include at least 10 subjects (up to 14 if needed to reach the 200 necessary data points to meet the ISO 80601-2-61:2017).
  Per FDA guidance, at least 2, or 15% of the subjects will have dark skin
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2021-12-16 (Actual); Study Completion 2021-12-16 (Actual)

PRIMARY OUTCOMES:
To obtain a reading from the Respiree device that corresponds to the associated blood sample or a reference oximeter. | 1 hour per subject
  The number of subjects and the number of comparisons (paired pulse oximeter readings and arterial saturation values) is determined by current FDA guidance requirements. This is a minimum of 200 data points and 10 subjects. In the course of this type of study, some subjects may drop out, some readings can be lost due to motion or other interference and occasionally some do not consent.

CONTACTS AND LOCATIONS:
Locations (1):
- Hypoxia Research Laboratory, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No